CLINICAL TRIAL: NCT05756010
Title: Effect of Forward Head Correction on EMG Activity of Masticatory and Cervical Muscles in Patients With Temporomandibular Disorder
Brief Title: Effect of Forward Head Correction on EMG of Masticatory Muscles in Patients With TMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Rami Abbas, Associate prof of physical therapy, Beirut Arab University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tempromandibular disorder TMD
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Temporomandibular Disorder
Keywords: TMJ pain; EMG activity; cervical pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): The program consisted of two strengthening (deep cervical flexors and shoulder retractors) and two stretchings (cervical extensors and pectoral muscles) exercises based on Harman and Mostafa et al's approach.
  Interventions: Device: EMG
- conrol group (Sham Comparator): General exercises
  Interventions: Device: EMG

INTERVENTIONS:
Device: EMG — The program consisted of two strengthening (deep cervical flexors and shoulder retractors) and two stretchings (cervical extensors and pectoral muscles) exercises
  Other Names: Forward head correction

SUMMARY:
This study aims to investigate the effects of forward head correction exercises on EMG of masticatory and cervical muscles in patients with temporomandibular disorder. The study's design will be double-blinded, randomized controlled trial. Patients suffering from TMD will be included in the program. The participants will allocate to one of two groups at random: the experimental group will perform a program consisting of two strengthening exercises (deep cervical flexors and shoulder retractors) and two stretchings (cervical extensors and pectoral muscles) and the control group will receive only neck flexion exercise.. This exercise program will be repeated 4 times per week for 10 weeks, and each session lasted for 30 minutes. The muscle activity EMG of masseter, temporalis, splenius, upper trapezius, and SCM will be measured pre and post-assessment using a biopic data acquisition system.

DETAILED DESCRIPTION:
1- EMG activity: Electrodes will be placed on the muscle belly parallel to the direction of muscle fibers. The distance between the two electrodes was 2 cm. The subjects will instructs to complete maximum voluntary contraction (MVC) by clenching the teeth for 3 s and repeating twice. The average of the two trials of MVC was used for further analysis.

1. To test the masseter and temporalis muscles: The subjects will be seated on a stable chair and will be instructed to tightly bite a cotton roll 10 mm thick as much as possible.
2. To test splenius muscle: the subjects will be seated on a stable chair and the examiner resist head extension.
3. To test the upper trapezius muscle: The subjects will be seated on a stable chair with the head side bent to the opposite side of the tested muscle; the examiner resist head side bending and shoulder elevation.
4. To test the sternocleidomastoid muscle: The subjects will be placed in a supine position and the examiner resisted the movement of cervical flexion by lifting the head from the table, with the chin depressed and approximated toward the sternum.

2. Measurement of TMJ range of motion. An 11 cm plastic ruler marked in millimeters measured TMJ opening range of motion "Opening. The subject will be instructed to open his mouth as wide as possible without causing pain or discomfort. The rater will measured the intercisal distance by placing one end of the ruler against the incise edge of one of the central incisors, and the other end against the incise edge of the opposing maxillary incisor." TMJ ROM measurements will be taken once for all patients before subdividing into groups and then after treatment intervention methods.

3-Use of the Fonseca's questionnaire to assess the prevalence and severity of temporomandibular disorders The Fonseca's questionnaire which considered to be valid and reliable for collecting a large quantity of information in a relatively short period and at low cost, it was easy to understand and had almost no influence from the examiner.

-intervention program: The program consisted of two strengthening (deep cervical flexors and shoulder retractors) and two stretchings (cervical extensors and pectoral muscles) exercises based on Harman and Mostafa et al's approach..

ELIGIBILITY:
Inclusion Criteria:

* Men and women/aged between 18-40/ patients suffer from TMJ disorder/ no other treatment such as medications, physical therapy, and joint injections in the past 2 weeks

Exclusion Criteria:

* Previous history of TMG subluxation or dislocation that may interfere with the opening of the mouth/ Neck pain which may affect the head and neck posture/ Head or neck trauma/.Class II or III malocclusion/ posture disorder caused by abnormal curvature of the spine; rheumatic disease; hemorrhagic disease, etc.;/ Lateral deviation of the mandible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-29 (Estimated)

PRIMARY OUTCOMES:
EMG activity | 10 weeks
  Electrodes will placed on the muscle belly parallel to the direction of muscle fibers. The distance between the two electrodes was 2 cm. The subjects will instructed to complete maximum voluntary contraction (MVC) of clenching the teeth for a period of 3 s and repeated twice. The average of the two trials of MVC will used for further analysis. target muscles include masseter , temporalis, splenius, upper trapezius and sternocleidomastoid muscles.

SECONDARY OUTCOMES:
Measurement of TMJ range of motion. | 10 weeks
  The subject will instructed to open his mouth as wide as possible without causing pain or discomfort. The rater will measured the intercisal distance by placing one end of the ruler against the incise edge of one of the central incisors, and the other end against the incise edge of the opposing maxillary incisor." TMJ ROM measurements will be taken once for all patients before subdividing into groups and then after treatment intervention methods.
Fonseca's questionnaire | 10 weeks
  assess the prevalence and severity of temporomandibular disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed ElMelhat, Professor, Study Chair — Assistant Prof of Physical Therapy
Locations (1):
- Physical therapy outpatient clinic, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Any study records that identify patient will be kept confidential. The records from the participation may be reviewed by people responsible for making sure that research is done properly, including members of the BAU Institutional Review Board. All of these people are required to keep their identities confidential. Otherwise, records that identify patients will be available only to people working on the study.
  • We will use a code of numbers and alphabets rather than participants' names on data sheets, keeping records in a safe place.

REFERENCES:
- [Background] Kim DH, Kim CJ, Son SM. Neck Pain in Adults with Forward Head Posture: Effects of Craniovertebral Angle and Cervical Range of Motion. Osong Public Health Res Perspect. 2018 Dec;9(6):309-313. doi: 10.24171/j.phrp.2018.9.6.04. PMID 30584494
- [Background] Ballenberger N, von Piekartz H, Paris-Alemany A, La Touche R, Angulo-Diaz-Parreno S. Influence of different upper cervical positions on electromyography activity of the masticatory muscles. J Manipulative Physiol Ther. 2012 May;35(4):308-18. doi: 10.1016/j.jmpt.2012.04.020. PMID 22632591
- [Background] Wang MQ, He JJ, Wang K, Svensson P. Influence of changing occlusal support on jaw-closing muscle electromyographic activity in healthy men and women. Acta Odontol Scand. 2009;67(3):187-92. doi: 10.1080/00016350902794800. PMID 19291503
- [Background] Yao Y, Cai B, Fan S, Yang HX, Zhang YX, Xu LL. The association between forward head posture and masticatory muscle pressure pain thresholds in patients with temporomandibular joint dissorders: a cross-sectional observational study. Clin Oral Investig. 2023 Jan;27(1):353-360. doi: 10.1007/s00784-022-04739-9. Epub 2022 Oct 14. PMID 36241923
- [Background] Xu L, Zhang L, Lu J, Fan S, Cai B, Dai K. Head and neck posture influences masticatory muscle electromyographic amplitude in healthy subjects and patients with temporomandibular disorder: a preliminary study. Ann Palliat Med. 2021 Mar;10(3):2880-2888. doi: 10.21037/apm-20-1850. Epub 2021 Mar 3. PMID 33691457
- [Background] Berni KC, Dibai-Filho AV, Pires PF, Rodrigues-Bigaton D. Accuracy of the surface electromyography RMS processing for the diagnosis of myogenous temporomandibular disorder. J Electromyogr Kinesiol. 2015 Aug;25(4):596-602. doi: 10.1016/j.jelekin.2015.05.004. Epub 2015 May 27. PMID 26054969
- [Background] Tecco S, Tete S, D'Attilio M, Perillo L, Festa F. Surface electromyographic patterns of masticatory, neck, and trunk muscles in temporomandibular joint dysfunction patients undergoing anterior repositioning splint therapy. Eur J Orthod. 2008 Dec;30(6):592-7. doi: 10.1093/ejo/cjn052. Epub 2008 Nov 5. PMID 18990679
- [Background] Chaves TC, Dos Santos Aguiar A, Felicio LR, Greghi SM, Hallak Regalo SC, Bevilaqua-Grossi D. Electromyographic ratio of masseter and anterior temporalis muscles in children with and without temporomandibular disorders. Int J Pediatr Otorhinolaryngol. 2017 Jun;97:35-41. doi: 10.1016/j.ijporl.2017.03.022. Epub 2017 Mar 18. PMID 28483248
- [Background] Cuenca-Martinez F, Herranz-Gomez A, Madronero-Miguel B, Reina-Varona A, La Touche R, Angulo-Diaz-Parreno S, Pardo-Montero J, Del Corral T, Lopez-de-Uralde-Villanueva I. Craniocervical and Cervical Spine Features of Patients with Temporomandibular Disorders: A Systematic Review and Meta-Analysis of Observational Studies. J Clin Med. 2020 Aug 30;9(9):2806. doi: 10.3390/jcm9092806. PMID 32872670